CLINICAL TRIAL: NCT00233207
Title: Acute Lung Injury Clinical Trials Incubator Unit
Brief Title: IC14 Antibodies to Treat Individuals With Acute Lung Injury
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Unable to meet enrollment number to complete study, study stopped June 30, 2007
Sponsor: University of Washington (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: 328; P50HL073996 (NIH)
Record Dates: First submitted 2005-10-03; First posted 2005-10-05 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2007-12

CONDITIONS: Respiratory Distress Syndrome, Adult; Lung Diseases
MeSH Terms: conditions — Respiratory Distress Syndrome; Lung Diseases

INTERVENTIONS:
Drug: IC14

SUMMARY:
This is a phase II, randomized, double-blind, placebo-controlled, safety and efficacy study of a recombinant chimeric monoclonal antibody against CD14 (IC14) in hospitalized patients with acute lung injury (ALI).

DETAILED DESCRIPTION:
BACKGROUND:

This study will use IC14, a recombinant chimeric monoclonal antibody (mAb) recognizing CD14, to block CD14 medicated cellular activation in patients with sepsis-induced ALI. Research results of antibody interaction with CD14 suggest that CD14 has a central role in the recognition of bacterial products and the induction of innate immune responses. Although beneficial, when this response is combined with a component of alveolar stretch it may induce an exaggerated response that can be harmful. This study will implement strategies to block CD14-mediated cellular activation and will evaluate whether this strategy has a beneficial effect in reducing alveolar inflammatory response, mechanical ventilation days, multiple organ failure, and severity of organ dysfunction in patients with sepsis-induced ALI.

DESIGN NARRATIVE:

The primary outcome of this study will be alveolar lavage concentrations of interleukin-8 that will be measured post-treatment at Days 2 and 3, and Days 6 to 8.

The key secondary outcomes of this study will be: 1) Worst Murray Lung Injury Score (measured at Days 1 through 7, and Day 28); 2) Worst Multiple Organ Dysfunction (MOD) Score (Marshall) (measured at Days 1 through 7, and Day 28); 3) Infections-nosocomial and/or surgical site infections (measured at Day 28); 4) Ventilator-free days (measured at Day 28); and 5) Mortality (measured at Day 28).

ELIGIBILITY:
Inclusion Criteria:

* Presence of ALI, defined as the following:

  1. Acute onset (less than 28 days from study entry)
  2. PaO2/FiO2 of less than 300
  3. Bilateral infiltrates consistent with pulmonary edema on frontal chest radiograph (infiltrates may be patchy, diffuse, homogeneous, or asymmetric)
  4. Requirement for positive pressure ventilation via endotracheal tube
  5. No clinical evidence of left atrial hypertension
* Clinical indication for antimicrobial therapy at the time of randomization
* Anticipated duration of mechanical ventilation greater than 48 hours

Exclusion Criteria:

* Treatment with a drug or device within 30 days prior to study entry that has not received regulatory approval at the time of study entry
* Does not meet safety criteria for bronchoscopic alveolar lavage either at baseline or is anticipated to be too high a risk for lavage on Day 1 of the study
* Intubation for cardiopulmonary arrest
* Intubation for status asthmaticus, pulmonary embolus, or myocardia infarction
* Anticipated survival less than 48 hours from intubation
* Anticipated survival less than 28 days due to pre-existing medical condition

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2005-09; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Alveolar lavage concentrations of interleukin-8 (measured post-treatment at Days 2, 3, 6, 7, and 8)

SECONDARY OUTCOMES:
Worst Murray Lung Injury Score
Worst Multiple Organ Dysfunction (MOD) Score (Marshall) (measured at Days 1 through 7, and Day 28)
Infections-nosocomial and/or surgical site infections
Ventilator-free days
Mortality (measured at Day 28)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Neff, MD, Study Chair — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States